CLINICAL TRIAL: NCT04515498
Title: A Prospective Clinical Study of the Ability of the CloudCath System to Detect Peritonitis During In-home Peritoneal Dialysis
Brief Title: A Prospective Clinical Study of the CloudCath System During In-home Peritoneal Dialysis
Acronym: CATCH
Status: Completed | Type: Observational
Sponsor: CloudCath (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-P-001
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Peritoneal Dialysis-associated Peritonitis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- CloudCath System: Patients with End Stage Renal Disease (ESRD) currently using home peritoneal dialysis
  Interventions: Device: CloudCath Monitoring System

INTERVENTIONS:
Device: CloudCath Monitoring System — The CloudCath Monitoring System will analyze effluent dialysate for changes associated with peritonitis.

SUMMARY:
This study aims to determine if the CloudCath device can detect infections related to peritoneal dialysis (peritonitis) as fast or faster than the current standard methods used by patients and doctors to detect such infections.

DETAILED DESCRIPTION:
This study will evaluate the safety and effectiveness of the CloudCath System to detect the onset of peritonitis as compared to standard of care.

Study Participants will connect the CloudCath System to their home peritoneal dialysis unit and the CloudCath System will analyze the effluent dialysis solution for changes associated with peritonitis. The notification capability of the CloudCath System will be deactivated for this study so that neither Study Participants nor Study Investigators will be aware of the device measurements.

Following enrollment, Study Participants will use the CloudCath System for 12 continuous months.

ELIGIBILITY:
Key Inclusion Criteria:

* currently using peritoneal dialysis
* provides informed consent
* willing to comply with the requirements of the study
* has cellular data coverage at home

Key Exclusion Criteria:

* active or history of cancer requiring chemotherapy within prior 6 months
* signs or symptoms of an active infection within 14 days prior to enrollment
* peritonitis diagnosis within 30 days prior to enrollment
* participating in another investigational device or drug study that may potentially affect study results
* other medical, social or psychological problems that, in the opinion of the investigator, exclude the study participant from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients currently using home peritoneal dialysis.
Sampling Method: Non-Probability Sample
Enrollment: 243 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Time of peritonitis detection (vs lab measures) | through 12 months
  The time peritonitis is detected by the CloudCath System, as compared to time of laboratory evidence of peritonitis

SECONDARY OUTCOMES:
Time of peritonitis detection (vs clinical measures) | through 12 months
  The time peritonitis is detected by the CloudCath System, as compared to time of peritonitis detection by standard clinical means (ISPD guidelines)
Sensitivity and specificity of the CloudCath System detection of peritonitis | through 12 months
  Analysis of sensitivity and specificity of CloudCath System detection of peritonitis, as compared to diagnostic laboratory testing
Ability of study participants to use the CloudCath System as intended | through 12-months of study follow-up
  Device performance measure; ability to use as intended

OTHER OUTCOMES:
Sensitivity and specificity of the CloudCath System detection of peritonitis and the resolution of peritonitis | through 12 months
  Analysis of sensitivity and specificity of the detection of peritonitis and the detection of the resolution of peritonitis, as compared to diagnostic laboratory testing
Sensitivity and specificity of the CloudCath System detection of resolution of peritonitis | through 12 months
  Analysis of sensitivity and specificity of the resolution time of peritonitis

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Chertow, MD, Study Director — Stanford University
Locations (1):
- CloudCath Investigational Site, Lakewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No